CLINICAL TRIAL: NCT00266851
Title: AZMATICS: Azithromycin Asthma Trial In Community Settings
Brief Title: AZMATICS: AZithroMycin/Asthma Trial In Community Settings
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: American Academy of Family Physicians (Other); Dean Foundation (Other); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-2005-0258
Record Dates: First submitted 2005-12-15; First posted 2005-12-19 (Estimated); Results first posted 2019-09-06 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-07

CONDITIONS: Asthma
Keywords: Randomized clinical trial; Asthma; Adults; Azithromycin
MeSH Terms: conditions — Asthma | interventions — Azithromycin

STUDY DESIGN:
Intervention Model Description: 2 arms are randomized, placebo-controlled, double-blinded, 1 arm was added as an open-label observational cohort
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Azithromycin (Active Comparator): Active adjunctive treatment
  Interventions: Drug: Azithromycin
- Placebo (Placebo Comparator): Adjunctive placebo
  Interventions: Drug: Placebo
- Observational Cohort (Other): Eligible participants who declined randomization, offered enrollment in parallel, open-label azithromycin treatment arm
  Interventions: Drug: Azithromycin

INTERVENTIONS:
Drug: Azithromycin — 600 mg x 3 days, then 600 mg weekly x 11 weeks
  Other Names: Zithromax
  Arms: Azithromycin; Observational Cohort
Drug: Placebo — Matching placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the effectiveness of the azalide macrolide azithromycin in adults with persistent asthma.

Research Question: Will a 12-week treatment with the antibiotic, azithromycin, result in a statistically significant and clinically meaningful improvement in overall asthma symptoms and other patient-oriented asthma outcomes one year after initiation of treatment of adult primary care patients with asthma?

Experimental Design: The investigators propose a one-year randomized, placebo-controlled, blinded (investigator, patient, data collector, data analyst) trial of 12 weekly doses of azithromycin/placebo as adjunctive therapy (in addition to usual care) along with a parallel observational cohort who will participate 'open label' in 100 adult asthma patients recruited from practice-based research networks (e.g., Wisconsin Research and Education Network (WREN) and others). This "practical clinical trial" will (1) enroll a representative sample of asthma patients encountered in the practices of primary care physicians, (2) employ standard clinical trial methodology to ensure internally valid results and (3) measure outcomes important to patients, so that the results will be valid and applicable to the kinds of asthma patients encountered by family physicians and other primary care providers.

Active study sites -

* Wisconsin: Augusta, Cross Plains, La Crosse, Marshfield, Milwaukee, Madison,
* Mauston, Rice Lake, Tomah, Wausau
* Colorado: Monument
* Illinois: Peoria
* Nevada: Reno
* North Carolina: Granite Falls
* North Dakota: Minot
* Ohio: Cleveland, Berea
* Oklahoma: Ardmore, Claremore, Edmond, Lawton, Oklahoma City, Stroud, Tulsa, Weatherford
* Rhode Island: East Providence

DETAILED DESCRIPTION:
1.0 PROTOCOL SYNOPSIS

Approximately 100 eligible adult patients with physician-diagnosed asthma will either be randomized to 12-week treatment with azithromycin or an identical placebo, or join an observational open-label azithromycin cohort. Azithromycin is a widely marketed azalide antibiotic with an excellent safety profile. Azithromycin or placebo will be adjunctive therapy for usual asthma care. The following patient-reported data will be collected via Zoomerang™ (a commercially-available data collection tool) periodically until one year after randomization: (1) study medication adherence and side effects weekly until 12 weeks, (2) asthma control and exacerbations every 6 weeks until 12 months, and (3) asthma quality of life and asthma controller medication changes every 3 months until 12 months. The primary hypothesis is that azithromycin will significantly improve asthma control (decrease symptoms and medication use) by 3 months (end treatment) and the improvement will continue to 12 months (end study). The primary outcome variable is overall asthma symptoms. Secondary outcomes are asthma medication use, quality of life and exacerbations. We will examine the predictive value of baseline patient characteristics including age, sex, smoking, co-morbid respiratory diagnoses and degree of airflow limitation. We will also examine for any imbalances between study groups in controller medication use, other antibiotic prescriptions and acute respiratory illnesses during the one-year study period.

We will enroll subjects from the practices of Wisconsin Research and Education Network (WREN) members, UW Department of Family Medicine physicians, Dean Medical Center primary care physicians, and from other practice-based research networks (PBRNs), medical group practices and individual primary care practices throughout North America.

Patients with physician-diagnosed asthma aged 18 and older will be identified at point-of-service (office, urgent care, emergency room or hospital), by administrative data base review, or by physician recall. Most subjects will be the patients of study physicians. Other physicians in the group practice may refer subjects. Subjects also may be self-referred after responding to posters placed in the clinics. Some sites may elect to identify cases by medical record or database review, in which case only the personal physician may initiate patient contacts.

Treatment is azithromycin tablets, 600 milligrams orally once daily for 3 days, then 600 milligrams once weekly for an additional 11 weeks (total dose 8400 milligrams) or identical placebo, in addition to usual care for asthma.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and older (and at least 50 kg/110 pounds)

  * The lower weight limit was chosen to avoid exposure to greater than 12 mg/kg/day of azithromycin (a currently recommended dose for children)
  * We specify no upper age limit because asthma occurs throughout the age range and because asthma in the elderly is particularly severe and warrants inclusion.
* Physician-diagnosed asthma
* At the time of randomization, eligible subjects must either:

  * be having a documented asthma exacerbation OR
  * be reporting at least mild persistent asthma symptoms, as defined by GINA (Global Initiative for Asthma)
* Subjects must also have asthma symptoms for at least six months prior to randomization
* Documentation of objective evidence of reversible airway obstruction, either spontaneously or after treatment, is required prior to randomization. This requirement can be met by documentary evidence, within 2 years of randomization, of either:

  * a 12% or greater (and ≥200 mL) change in FEV1 OR
  * a 25% or greater (and >60 L/min) change in PEFR either spontaneously or as a result of treatment

Exclusion Criteria:

* Not English literate or without email and internet access
* Macrolide allergy
* Pregnancy or lactation
* Females of childbearing potential must agree to use an acceptable form of contraception during the treatment period
* Chronic use of macrolides, tetracyclines or quinolones Chronic use is defined as 4 or more weeks of continuous use within 6 months of randomization
* Asthma symptoms for less than 6 months prior to randomization Asthma symptoms must be present for at least 6 months to exclude patients without true chronic asthma
* Unstable asthma requiring immediate emergency care All patients with asthma exacerbations will receive usual urgent or emergency care for asthma and must be improving or stable in the judgment of the treating physician prior to being enrolled
* Specified co-morbidities likely to interfere with study assessments or follow up. Excluded comorbidities include:

  * cystic fibrosis
  * obstructive sleep apnea requiring CPAP
  * cardiomyopathy
  * congestive heart failure
  * terminal cancer
  * alcohol or other drug abuse
  * or any other serious medical condition that, in the opinion of the study physician, would seriously interfere with or preclude assessment of study outcomes or completion of study assessments
* Specified medical conditions for which macrolide administration may possibly be hazardous
* Patients with acute or chronic hepatitis, cirrhosis or other liver disease, chronic kidney disease, or history of prolonged cardiac repolarization and QT interval or torsades de pointes, are excluded
* Specified medications for which close monitoring has been recommended in the setting of macrolide administration Patients taking digoxin, theophylline, warfarin, ergotamine or dihydroergotamine, triazolam, carbamazepine, cyclosporine, hexobarbital or phenytoin are excluded.

  * If any of these medications are started after randomization and before completion of the 12-week treatment phase, study medication will be discontinued and the patient may remain in the study.

The intent of this protocol is to enroll a broadly generalizable sample of adult patients with physician-diagnosed asthma, either stable persistent or in exacerbation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2006-01; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David L Hahn, MD, MS, Principal Investigator — Wisconsin Research and Education Network (WREN)
Locations (5):
- United States (5):
  - ANSR, Peoria, Illinois
  - AAFP National Research Network, Kansas City, Kansas
  - RAP - Cleveland Clinic, Cleveland, Ohio
  - University of Oklahoma Health Sciences Center (OUHSC) and Oklahoma Physicians Resource/Research Network (OKPRN), Oklahoma City, Oklahoma
  - Wisconsin Research and Education Network (WREN), Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hahn DL, Plane MB. Feasibility of a practical clinical trial for asthma conducted in primary care. J Am Board Fam Pract. 2004 May-Jun;17(3):190-5. doi: 10.3122/jabfm.17.3.190. PMID 15226283
- [Background] Hahn DL. Treatment of Chlamydia pneumoniae infection in adult asthma: a before-after trial. J Fam Pract. 1995 Oct;41(4):345-51. PMID 7561707
- [Background] Hahn DL. Chlamydia pneumoniae, asthma, and COPD: what is the evidence? Ann Allergy Asthma Immunol. 1999 Oct;83(4):271-88, 291; quiz 291-2. doi: 10.1016/S1081-1206(10)62666-X. PMID 10541419
- [Background] Hahn DL, Plane MB, Mahdi OS, Byrne GI. Secondary outcomes of a pilot randomized trial of azithromycin treatment for asthma. PLoS Clin Trials. 2006 Jun;1(2):e11. doi: 10.1371/journal.pctr.0010011. Epub 2006 Jun 30. PMID 16871333
- [Result] Hahn DL, Grasmick M, Hetzel S, Yale S; AZMATICS (AZithroMycin-Asthma Trial In Community Settings) Study Group. Azithromycin for bronchial asthma in adults: an effectiveness trial. J Am Board Fam Med. 2012 Jul-Aug;25(4):442-59. doi: 10.3122/jabfm.2012.04.110309. PMID 22773713
- See also: Patient perspective/literature review — http://www.asthmastory.com
- See also: Book that reviews the topic of infection as a treatable cause for asthma — https://www.peoplespharmacy.com/store/books/a-cure-for-asthma-what-your-doctor-isnt-telling-you-and-why/

RESULTS

PARTICIPANT FLOW:
Groups:
- Observational Cohort: Eligible participants that declined randomization were offered enrollment in open-label, azithromycin treatment arm
Period: Overall Study
Arm/Group | Placebo | Azithromycin | Observational Cohort
Started | 37 | 38 | 22
Completed 3 Month Follow up | 26 | 22 | 15
Completed 6 Month Follow up | 27 | 22 | 17
Completed 9 Month Follow up | 22 | 23 | 15
Completed 12 Month Follow up | 25 | 19 | 13
Completed (All participants received the intervention or participated in the open-label arm completed study.) | 37 | 38 | 22
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: all participants who received study intervention or observation
Groups:
- Observational Cohort: Eligible participants who declined randomization were offered enrollment in an observational open-label azithromycin arm
- Total: Total of all reporting groups
Arm/Group | Placebo | Azithromycin | Observational Cohort | Total
Number analyzed (Participants) | 37 | 38 | 22 | 97
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.4 (14.2) | 45.7 (15.5) | 45.4 (15.2) | 46.3 (14.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 27 | 10 | 61
  Male | 13 | 11 | 12 | 36
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 33 | 36 | 18 | 87
  Race: Unknown | 4 | 2 | 4 | 10
Region of Enrollment [Number; unit: participants]
  United States | 37 | 38 | 22 | 97
Smoking Status [Count of Participants; unit: Participants]
  Never | 13 | 20 | 16 | 49
  Former | 19 | 12 | 6 | 37
  Current | 5 | 6 | 0 | 11
Education [Median (Full Range); unit: years] | 15 [10 to 20] | 14 [12 to 22] | 17 [12 to 25] | 15 [10 to 25]
Chronic Sinusitis [Count of Participants; unit: Participants] | 11 | 14 | 19 | 44
Allergy Tested [Count of Participants; unit: Participants] — Population: Not all participants were allergy tested, this was a physician decision
  Participants
    Negative: number analyzed (Participants) | 18 | 18 | 19 | 55
    Negative | 2 | 1 | 6 | 9
    Positive for 1-3 positive: number analyzed (Participants) | 18 | 18 | 19 | 55
    Positive for 1-3 positive | 4 | 3 | 8 | 15
    Positive for equal to or greater than 4: number analyzed (Participants) | 18 | 18 | 19 | 55
    Positive for equal to or greater than 4 | 12 | 14 | 5 | 31
Infectious Asthma [Count of Participants; unit: Participants] — History showed first asthma symptoms began after an acute respiratory illness.
  Participants | 6 | 17 | 13 | 36
Exacerbations [Count of Participants; unit: Participants] — within the previous 2 years
  Participants
    Hospitalized | 0 | 2 | 4 | 6
    Emergency Visit | 14 | 19 | 9 | 42
    Steroid burst | 22 | 24 | 13 | 59
Baseline Asthma Severity [Count of Participants; unit: Participants] — Day: mild is greater than or equal to 2 days/week to less than daily; moderate is greater than or equal to 1 per day to less than continuous; severe is continuous.
  Night: mild is greater than or equal to 2 per month to 1 per week; moderate is is greater than or equal to 1 per week to 1 per night; severe is is greater than or equal to 1 per night.
  Participants
    Day Symptom Frequency: Mild to Moderate | 35 | 34 | 15 | 84
    Day Symptom Frequency: Severe | 2 | 4 | 7 | 13
    Night Symptom Frequency: Mild to Moderate | 33 | 33 | 15 | 81
    Night Symptom Frequency: Severe | 4 | 5 | 7 | 16
Coexisting COPD [Count of Participants; unit: Participants] — Chronic Obstructive Pulmonary Disease
  Participants | 8 | 5 | 2 | 15
Lung Function, FEV [Mean (Standard Deviation); unit: liters in one second] — Forced expiratory volume (FEV) in 1 second Population: data was unable to be collected from all participants
  liters in one second
    number analyzed (Participants) | 19 | 19 | 7 | 45
    (all) | 2.35 (1.31) | 2.33 (1.05) | 2.48 (1.19) | 2.36 (1.16)
Lung Function, PEFR [Mean (Standard Deviation); unit: liters per min] — peak expiratory flow rate Population: data was unable to be collected from all participants
  liters per min
    number analyzed (Participants) | 24 | 26 | 18 | 68
    (all) | 251 (105) | 273 (109) | 300 (105) | 272 (107)
Controller Medication [Count of Participants; unit: Participants]
  Inhaled Corticosteroid | 30 | 24 | 18 | 72
  Long-Acting Bronchodilator | 26 | 14 | 15 | 55
  Leukotriene Inhibitor | 8 | 9 | 6 | 23
  Oral Prednisone | 4 | 2 | 1 | 7
Baseline Asthma Measures [Mean (Standard Deviation); unit: scores on a scale] — * Asthma symptom scores (0 is none, 1 is mild, 2 is moderate, 3 is severe, 4 is worst ever)
  * AQL (Juniper AQL questionnaire), scored on a scale of 1-7 where higher numbers indicate improved quality of life.
  * Asthma control (mini-Juniper Asthma Control Questionnaire, without pulmonary function), scored on a scale of 0-6 where 0 is no impairment and 6 is maximum impairment.
  scores on a scale
    Overall Asthma Symptoms | 1.48 (0.94) | 1.42 (0.77) | 2.06 (0.73) | 1.57 (0.86)
    Asthma Quality of Life | 4.97 (1.28) | 4.98 (1.27) | 4.12 (1.29) | 4.79 (1.31)
    Asthma Control | 1.56 (1.02) | 1.75 (0.93) | 2.26 (1.35) | 1.78 (1.08)
Participant Age at Asthma Diagnosis [Mean (Full Range); unit: years] | 24 [0 to 59] | 24 [0 to 58] | 28 [11 to 59] | 25 [0 to 59]

OUTCOME MEASURES:

1. Primary Outcome: Change in Overall Asthma Symptoms From Baseline
Description: 5-point scale: 0=none, 1=mild, 2=moderate, 3=severe, 4=worst ever, the lower scores indicate improvement in asthma symptoms
Time Frame: Within the past 24 hours; measured every 1.5 months for one year
Population: All participants did not adhere to follow-up schedule
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Observational Cohort: Eligible Participants who declined randomization were offered enrollment in a parallel open-label observational treatment arm
Arm/Group | Placebo | Azithromycin | Observational Cohort
Number analyzed (Participants) | 37 | 38 | 22
units on a scale
  Change from Baseline to Week 6: number analyzed (Participants) | 30 | 33 | 16
  Change from Baseline to Week 6 | -0.60 (1.07) | -0.15 (0.83) | -0.88 (0.81)
  Change from Baseline to Week 12: number analyzed (Participants) | 23 | 32 | 16
  Change from Baseline to Week 12 | -0.48 (1.16) | -0.31 (0.74) | -1.0 (1.37)
  Change from Baseline to Week 18: number analyzed (Participants) | 27 | 31 | 16
  Change from Baseline to Week 18 | -0.15 (1.13) | 0.10 (0.75) | -0.94 (1.12)
  Change from Baseline to Week 24: number analyzed (Participants) | 25 | 30 | 17
  Change from Baseline to Week 24 | -0.08 (0.95) | -0.10 (0.96) | -1.0 (1.17)
  Change from Baseline to Week 30: number analyzed (Participants) | 22 | 29 | 16
  Change from Baseline to Week 30 | -0.05 (1.09) | -0.34 (1.01) | -0.81 (1.17)
  Change from Baseline to Week 36: number analyzed (Participants) | 24 | 27 | 15
  Change from Baseline to Week 36 | -0.21 (1.14) | -0.22 (0.70) | -1.27 (0.70)
  Change from Baseline to Week 42: number analyzed (Participants) | 23 | 25 | 14
  Change from Baseline to Week 42 | -0.04 (0.88) | -0.12 (0.93) | -1.21 (0.70)
  Change from Baseline to Week 48: number analyzed (Participants) | 20 | 29 | 13
  Change from Baseline to Week 48 | -0.10 (1.07) | -0.07 (0.88) | -1.07 (0.95)

2. Secondary Outcome: Change in Asthma Control Over Baseline
Description: Mini-Juniper Asthma Control Questionnaire without pulmonary function. This is a 6-item survey scored on a 7 point scale where 0 is none, or no symptoms and 6 is severe or symptoms all of the time. Answers are averaged for a final score of 0-6. Data are reported as a change from baseline.
Time Frame: Within the past week; every 3 months
Population: All participants did not adhere to follow-up schedule
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- Observational Cohort: Eligible participants who declined randomization were offered enrollment in an open-label observational treatment arm.
Arm/Group | Placebo | Azithromycin | Observational Cohort
Number analyzed (Participants) | 37 | 38 | 22
scores on a scale
  Change from Baseline to Week 6: number analyzed (Participants) | 30 | 33 | 16
  Change from Baseline to Week 6 | -0.37 (0.88) | -0.46 (0.60) | -1.24 (1.14)
  Change from Baseline to Week 12: number analyzed (Participants) | 23 | 32 | 16
  Change from Baseline to Week 12 | -0.41 (1.01) | -0.40 (0.80) | -1.38 (1.87)
  Change from Baseline to Week 18: number analyzed (Participants) | 27 | 31 | 16
  Change from Baseline to Week 18 | -0.40 (1.05) | -0.28 (0.88) | -1.18 (1.53)
  Change from Baseline to Week 24: number analyzed (Participants) | 25 | 30 | 17
  Change from Baseline to Week 24 | -0.37 (1.12) | -0.34 (1.03) | -1.35 (1.69)
  Change from Baseline to Week 30: number analyzed (Participants) | 22 | 29 | 16
  Change from Baseline to Week 30 | -0.25 (1.22) | -0.56 (0.81) | -1.04 (1.38)
  Change from Baseline to Week 36: number analyzed (Participants) | 24 | 27 | 15
  Change from Baseline to Week 36 | -0.39 (1.00) | -0.39 (0.79) | -1.63 (1.41)
  Change from Baseline to Week 42: number analyzed (Participants) | 23 | 25 | 14
  Change from Baseline to Week 42 | -0.22 (1.32) | -0.38 (0.72) | -1.42 (1.41)
  Change from Baseline to Week 48: number analyzed (Participants) | 20 | 29 | 13
  Change from Baseline to Week 48 | -0.45 (1.00) | -0.34 (0.88) | -1.08 (1.20)

3. Secondary Outcome: Change is Asthma-specific Quality-of-Life (AQL)
Description: Juniper Asthma Quality of Life Questionnaire is a 32-item survey, recall of the past 2 weeks, scored on a 7 point Likert scale where 1 is severely impaired, and 7 is not impaired at all. Scores are averaged for a final range of 1-7. Change from Baseline is reported here.
Time Frame: Within the past 2 weeks; every three months
Population: All participants did not adhere to follow-up schedule
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Azithromycin | Observational Cohort
Number analyzed (Participants) | 37 | 38 | 22
score on a scale
  Change from Baseline to Week 12: number analyzed (Participants) | 22 | 26 | 15
  Change from Baseline to Week 12 | 0.50 (0.95) | 0.67 (1.10) | 1.54 (1.91)
  Change from Baseline to Week 24: number analyzed (Participants) | 22 | 27 | 17
  Change from Baseline to Week 24 | 0.31 (1.36) | 0.49 (1.11) | 1.36 (1.75)
  Change from Baseline to Week 36: number analyzed (Participants) | 23 | 22 | 15
  Change from Baseline to Week 36 | 0.23 (1.02) | 0.58 (1.04) | 2.05 (1.40)
  Change from Baseline to Week 48: number analyzed (Participants) | 19 | 25 | 13
  Change from Baseline to Week 48 | 0.40 (1.33) | 0.50 (1.10) | 1.70 (1.42)

4. Secondary Outcome: Asthma Exacerbations
Description: A steroid burst, an unscheduled or emergency visit and/or a hospitalization for asthma, reported at Weeks 0, 6, 12, 18, 24, 30, 36, 42, 48, and any time during follow up.
Time Frame: up to 12 months
Population: This study was not powered to detect significant differences in exacerbation frequency.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Randomized placebo
- Azithromycin: Randomized azithromycin
- Open-Label Azithromycin: Eligible participants who declined randomization were offered enrollment in an open-label observational treatment arm.
Arm/Group | Placebo | Azithromycin | Open-Label Azithromycin
Number analyzed (Participants) | 37 | 38 | 22
Participants
  Week 0: number analyzed (Participants) | 33 | 36 | 18
  Week 0 | 9 | 9 | 6
  Week 6: number analyzed (Participants) | 32 | 33 | 19
  Week 6 | 9 | 6 | 3
  Week 12: number analyzed (Participants) | 25 | 32 | 18
  Week 12 | 3 | 6 | 4
  Week 18: number analyzed (Participants) | 28 | 31 | 16
  Week 18 | 5 | 6 | 3
  Week 24: number analyzed (Participants) | 26 | 26 | 12
  Week 24 | 6 | 4 | 5
  Week 30: number analyzed (Participants) | 23 | 29 | 16
  Week 30 | 4 | 6 | 6
  Week 36: number analyzed (Participants) | 26 | 27 | 15
  Week 36 | 5 | 7 | 2
  Week 48: number analyzed (Participants) | 22 | 29 | 13
  Week 48 | 5 | 7 | 2
  At any time during follow up: number analyzed (Participants) | 33 | 36 | 19
  At any time during follow up | 15 | 20 | 10

ADVERSE EVENTS:
Time Frame: up to 12 weeks
Groups:
- Observational Cohort: Eligible participants who refused randomization were offered enrollment in an open-label azithromycin arm
Arm/Group | Placebo | Azithromycin | Observational Cohort
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/38 | 0/22
Serious Adverse Events (participants affected / at risk) | 1/37 | 0/38 | 0/22
Other Adverse Events (participants affected / at risk) | 7/34 | 16/35 | 14/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=37) | Azithromycin (N=38) | Observational Cohort (N=22)
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=34) | Azithromycin (N=35) | Observational Cohort (N=20)
Nausea (Gastrointestinal disorders) | 3 | 10 | 8
Vomiting (Gastrointestinal disorders) | 2 | 2 | 2
Stomach Pain (General disorders) | 4 | 11 | 11
Diarrhea (Gastrointestinal disorders) | 5 | 12 | 11
Rash (Skin and subcutaneous tissue disorders) | 1 | 3 | 4
Swelling (General disorders) | 0 | 2 | 2
Hearing Loss (Ear and labyrinth disorders) | 2 | 1 | 1
Vaginal Candidasis (Reproductive system and breast disorders) | 3 | 4 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No